CLINICAL TRIAL: NCT04640454
Title: Assessment of Nipple Sparing Mastectomy as a Treatment Option for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 13-27-10
Record Dates: First submitted 2020-11-05; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; mastectomy; breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: nipple sparing mastectomy — The investigators categorized the incisions into radial, inframammary, and periareolar incisions with planned reconstruction types; direct to implant (DTI), transversus rectus abdominis myocutaneous (TRAM) flap, latissimus dorsi myocutaneous (LD) flap, or LD with implant.

SUMMARY:
Nipple-sparing mastectomy (NSM) with immediate breast reconstruction (IBR) is a form of mastectomy that achieves optimal disease control and facilitates reconstruction. The study aimed to assess the oncological safety and aesthetic outcomes of nipple-sparing mastectomy and immediate breast reconstruction.

35 female patients with breast cancer were included in the study. The investigators categorized the incisions into radial, inframammary, and periareolar incisions with planned reconstruction types; direct to implant (DTI), transversus rectus abdominis myocutaneous (TRAM) flap, latissimus dorsi myocutaneous (LD) flap, or LD with implant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ductal in situ carcinoma or infiltrating ductal carcinoma with a tumor diameter up to 3 cm
* Distance of the tumor from the nipple ≥ 2 cm
* Cancer or microcalcifications not localized in the central field.
* No blood secretions or other (nipple-areola complex) NAC disturbances
* Absence of skin involvement
* Indication to mastectomy for multifocal or diffuse microcalcifications
* Negative intraoperative assessment of NAC-bottom

Exclusion Criteria:

* Tumor or microcalcifications localized in the central quadrant or in the retroareolar region
* Blood secretions or other NAC alterations
* Positive intraoperative assessment of NAC-bottom
* Inflammatory carcinoma
* Paget's disease of the nipple

Ages: 28 Years to 68 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The mean age of the studied patients was 44.00±9.47 years old; the youngest patient was 28 years old and the oldest one was 68 years old, the majority of patients were 40-50 years of age (54%) As regard the patients' marital status; 31 patients were married constituting 88.57 % and only 4 (11.4 %) patients were single The main complaint of 25 of them (71.42%) was painless breast lump while 8 cases (22.85%) presented with local recurrence after previous breast conservative surgery and only two case (5.7%) presented by extensive mammographic calcifications on screening mammography
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
patients complications after nipple sparing mastectomy | 2017-2019
  Complete general examination, local examination of the skin, nipple and areola were done to determine whether the patients suffered from any complaints

SECONDARY OUTCOMES:
Aesthetic results assessed by Tzafetta et al scoring system | 2017-2019

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria faculty of medicine, Alexandria, Egypt